CLINICAL TRIAL: NCT04511273
Title: Does Mirabegron Have a Positive Impact on Sexual Function in Females With Overactive Bladder ?
Brief Title: Does Mirabegron Have a Positive Impact on Sexual Function in Females With Overactive Bladder
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Samer Morsy, Urology Consultant, Kasr El Aini Hospital
Other Study IDs: Cairo University Hospitals
Record Dates: First submitted 2020-08-08; First posted 2020-08-13 (Actual); Last update posted 2020-08-13 (Actual); Status verified 2020-08

CONDITIONS: Females With Overactive Bladder Symptoms, Urgency & Urge Incontinence
MeSH Terms: conditions — Urinary Incontinence, Urge

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: Follow up of female sexual function — Mirabegron 50mg once daily for treatment of overactive bladder symptoms

SUMMARY:
80 female patients evaluated for sexual function after receiving Mirabegron 50 mg once daily for 6 months for treatment of overactive bladder symptoms

DETAILED DESCRIPTION:
80 female patients evaluated for sexual function after receiving Mirabegron 50 mg once daily for 6 months for treatment of overactive bladder symptoms

ELIGIBILITY:
Inclusion Criteria:

* any female with overactive bladder symptoms, urgency and urgency incontinence

Exclusion Criteria:

* neurologic abnormalities
* Weak bladder contractility
* Diabetics

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Females with overactive bladder symptoms
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2020-10-01 (Estimated); Study Completion 2021-04-01 (Estimated)

PRIMARY OUTCOMES:
Sexual function evaluation after 6 months | 6 months
  Sexual function evaluation using female sexual function index FSFI